CLINICAL TRIAL: NCT03449615
Title: Isotopic Versus Magnetic Intraoperative Node Evaluation in Cutaneous Malignant Melanoma
Brief Title: Validation of Ferromagnetic Tracer in Melanoma Sentinel Node
Acronym: IMINEM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sociedad Española de Oncología Quirúrgica (Other)
Collaborators: Sysmex España (Industry)
Responsible Party: Principal Investigator, Antonio Piñero-Madrona, SEOQ Researcher, Sociedad Española de Oncología Quirúrgica
Other Study IDs: SEOQ-MEL001
Record Dates: First submitted 2018-02-17; First posted 2018-02-28 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Melanoma Stage; Sentinel Lymph Node
Keywords: Cutaneous melanoma; Sentinel node biopsy
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study has been designed to validate a non-radioactive method to identify the sentinel lymph node using a superparamagnetic iron-oxide (SPIO) tracer respect to the traditional isotopic method. Both methods are used in every included patient and each patient is its own control.

DETAILED DESCRIPTION:
* Injection of the isotopic tracer in standard form and in the usual preoperative period (hours-day).
* Identical injection in three-four punctures of 2 mL of Sienna+ ® and local massage of 5-10 minutes.
* Optional: colorant injection in standard form. Local massage of 5-10 minutes.
* After 20 minutes: transcutaneous measurement with SentiMag®
* Valuing territories (lymphoscintigraphy information?)
* Surgical identification measures:

  1. st with SentiMag®
  2. nd with gamma detection probe
* Ex vivo check and HRD record

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years of age),
* with diagnosis of cutaneous melanoma and
* in which SLNB is indicated as a staging method, and
* with cN0 result after clinical-echographic-cytohistological evaluation.

Exclusion Criteria:

* Previous treatment with systemic therapy.
* Recent previous surgery (<3 months) in the area susceptible of lymphatic drainage from the melanoma.
* Intolerance or hypersensitivity to iron or dextran compounds.
* Impossibility of use of radioisotope.
* Existence of pathology related to elevation of organic iron (hemosiderosis, hemochromatosis, iron deficiency anemia of metabolic or circulatory origin).
* Implantation of pacemakers or partially or totally metallic thoracic implants.
* Treatment with iron chelators (deferasirox, deferoxamine, ...).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with cutaneous malignant melanoma with indication for sentinel lymph node biopsy in staging.
Sampling Method: Non-Probability Sample
Enrollment: 186 (Estimated)
Dates: Start 2015-12-21 (Actual); Primary Completion 2018-05 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
SN detection | During surgery
  Detection of potential sentinel nodes using both methods (isotopic and ferromagnetic tracers). Máximum register of isotopic and ferromagnetic measurement will be the main criteria.

SECONDARY OUTCOMES:
SN agreement | During surgery
  Agreement in isotopic and ferromagnetic sentinel node identification. Measurement criteria will be coincidence in the same node (or nodes).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico Universitario "Virgen de la Arrixaca", Murcia, Spain